CLINICAL TRIAL: NCT05738096
Title: Trigeminal Evoked Responses to Improve Rhizotomy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Rhizotomy
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Trigeminal Neuralgia; Rhizotomy
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TGN patients (Experimental): Patients with TGN who will undergo rhizotomy surgery as the standard of care
  Interventions: Other: TSEP + rhizotomy surgery
- Healthy volunteers (Active Comparator): Healthy volunteers for whom TSEPS will be recorded in a lab setting
  Interventions: Other: TSEPs recording only

INTERVENTIONS:
Other: TSEP + rhizotomy surgery — TGN patients recruited for this study will already be undergoing percutaneous rhizotomy surgery. TSEPs will be measured at baseline prior to surgery. During the rhizotomy procedure, an electrode or balloon is placed through a metal sheath to then damage the nerve. A stylet is introduced to clear tissue from the sheath in preparation for the electrode or balloon. Prior to the final insertion of the RF electrode where the gasserian ganglion will be damaged, we will place a standard stereotactic EEG electrode (SEEG). Following damaging the nerve (clinical procedure), we will record again to measure differences in the TSEPs following cell body damage. The Neuralynx system will be used to record the potentials at 40 KHz.
  Arms: TGN patients
Other: TSEPs recording only — TSEPS will also be recorded from healthy controls in a lab setting; all procedures for the healthy controls will be non-invasive.
  Arms: Healthy volunteers

SUMMARY:
Trigeminal neuralgia (TGN) is a debilitating pain syndrome where electrical, shock- like jolts of pain affect the face. Trigeminal somatosensory evoked potentials (TSEPs) provide a promising modality for measuring the trigeminal sensory and nociceptive pathway by using peripheral stimulation of the trigeminal nerve (on the skin) and measuring low latency evoked potentials on the scalp (contralateral sensory cortex). While TSEPs have been measured in the past, it is not clear if implementing TSEPs into a routine neurosurgical rhizotomy procedure will be feasible. This is a prospective cohort study examining the feasibility of routinely performing TSEPs during rhizotomies for TGN.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or older
* Scheduled to undergo percutaneous rhizotomy for facial pain

Exclusion Criteria:

* For TGN: Facial pain of unclear origin (i.e. not clearly TGN pain) or Rhizotomy procedure canceled
* For Healthy control: Diagnosis or history of facial pain such as TMD or TGN, History of migraine, History of any functional pain disorder: fibromyalgia, IBS, CRPS or Recent chronic pain (within last month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 years
  total study procedure completion rate

SECONDARY OUTCOMES:
TSEPS peak to peak amplitude within TGN | 1 day
  difference in measured peak to peak amplitude between normal and TGN side
TSEPS latency within TGN | 1 day
  difference in measured TSEPS latency between normal and TGN side
TSEPS peak to peak amplitude between control and TGN patients | 1 day
  difference in measured peak to peak amplitude between healthy participants and TGN patients
TSEPS latency between control and TGN patients | 1 day
  difference in latency between healthy participants and TGN patients

CONTACTS AND LOCATIONS:
Overall Officials: David P Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States